CLINICAL TRIAL: NCT03387384
Title: Appropriateness of Aspirin Use in Medical Outpatients: A Multicenter, Observational Study
Brief Title: Appropriateness of Aspirin Use in Medical Outpatients
Acronym: ASSOS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, OGUZHAN CELIK, Faculty of Medicine, Department of Cardiology, M.D., Principal Investigator, Muğla Sıtkı Koçman University
Other Study IDs: MuglaSKU2
Record Dates: First submitted 2017-12-01; First posted 2018-01-02 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Primary Prevention of Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non-interventional study — Non-interventional study

SUMMARY:
This study aims to describe the demographic characteristics and current status of the aspirin use for primary and secondary prevention of cardiovascular diseases in a large, multicenter nationwide study

DETAILED DESCRIPTION:
Although the benefit of aspirin use for secondary prevention is well established, its role in the primary prevention of cardiovascular diseases remains controversial. Differences in primary prevention guidelines may lead to underuse of aspirin in high-risk patients and overuse in low-risk patients. This study aims to describe the demographic characteristics and current status of the aspirin use for primary and secondary prevention of cardiovascular diseases in a large, multicenter nationwide study. The ASSOS trial (Appropriateness of Aspirin Use in Medical Outpatients: A Multicenter, Observational Study) will be an observational, multicenter, and non-interventional study conducted in Turkey. Approximately 5000 patients will be enrolled in this non-interventional study. All the data will be collected at one point in time and current clinical practice will be evaluated.

The investigators will enroll all consecutive patients admitted to the outpatient cardiology clinics from January 30, 2018, through May 30, 2018, who were at least 18 years of age, provided written informed consent, and currently treated with aspirin (80-325 mg)within the last 30 days. Hospital-based cardiologists in public units will be invited to participate in the study. Patients will be stratified into 2 categories based on the presence or absence of atherosclerotic cardiovascular disease; secondary prevention group and primary prevention group, respectively. Appropriateness of aspirin use in primary prevention group will be evaluated according to the US Preventive Services Task Force (USPSTF) and European Society of Cardiology (ESC) guidelines. Physicians will complete a standardized survey form to collect information on patient clinical characteristics, cardiovascular risk factors, medical history, clinical examination, laboratory test results, and medications. Patients' risk factors for colorectal cancer and gastrointestinal bleeding will also be questioned.

ASSOS registry will be the largest and most comprehensive study in Turkey evaluating aspirin use. The results of this study will provide valuable information regarding the potential misuse of aspirin in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients using aspirin 18 years and older

Exclusion Criteria:

* Patients under 18 years of age
* Patients who do not want to participate in our study
* Patients who do not use aspirin

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All consecutive patients over the age of 18 using aspirin who presented to cardiology outpatient clinics will be screened
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-06-30 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-07-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of appropriate aspirin use in the primary prevention of cardiovascular diseases | 12 months
  Appropriate aspirin use will be defined with US Preventive Services Task Force (USPSTF).

CONTACTS AND LOCATIONS:
Locations (1):
- Mugla Sitki Kocman University Training and Research Hospital, Muğla, Turkey (Türkiye)

REFERENCES:
- [Derived] Celik O, Cil C, Ozlek B, Ozlek E, Dogan V, Basaran O, Demirci E, Bekar L, Kalcik M, Karaarslan O, Yetim M, Dogan T, Demir V, Kalkan S, Ozkan B, Hidayet S, Taylan G, Kucuksu Z, Celik Y, Efe SC, Aslan O, Biteker M. Design and rationale for the ASSOS study: Appropriateness of aspirin use in medical outpatients a multicenter and observational study. Anatol J Cardiol. 2018 Dec;20(6):354-362. doi: 10.14744/AnatolJCardiol.2018.47587. PMID 30504736